CLINICAL TRIAL: NCT05933837
Title: Association Between Troponin I Levels and Mortality Among Patients Undergoing Acute High-risk Abdominal Surgery - a Cohort Study
Brief Title: Troponin I Level and Mortality in Acute Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Tiffanie Bendtz Kanstrup, PhD, MD, Nordsjaellands Hospital
Other Study IDs: P-2020-507
Record Dates: First submitted 2023-06-20; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Myocardial Injury After Non-cardiac Surgery; Abdomen, Acute
Keywords: Myocardial injury after non-cardiac surgery; Abdomen, Acute; Troponin I; Myocardial Injury; Emergency surgery
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with MINS: Troponin I level equal to or above 59 ng/L
  Interventions: Diagnostic Test: Troponin I
- Patients without MINS: Troponin I level under 59 ng/L
  Interventions: Diagnostic Test: Troponin I

INTERVENTIONS:
Diagnostic Test: Troponin I — Measurements of plasma Troponin I 6-12 hours and on the first four postoperative days after surgery.

SUMMARY:
The goal of this prospective cohort study is to estimate the incidence of myocardial injury after non-cardiac surgery (MINS) in patients undergoing acute high-risk abdominal surgery.

MINS is defined as at least one increased single measurement of plasma troponin I (TnI). TnI-dynamic is defined as either two succeeding measurements of TnI > 59 ng/l with an increase/fall of more than 20%, or by one measurements of TnI > 59 ng/l with a succeeding measurement of TnI < 59 ng/l and a decrease of more than 50%.

Participants will have plasma TnI measured 6-12 hours postoperatively and on each of the following four postoperative days. Follow-up will be minimum one year after surgery.

The aim of the study is to determine:

* The incidence of MINS within the first four postoperative days
* The incidence of dynamic TnI changes
* The association between MINS and dynamic TnI changes respectively and all-course short-term mortality

DETAILED DESCRIPTION:
Gastrointestinal tract perforation, bowel ischemia and bowel obstruction are considered acute high-risk abdominal disorders, often requiring emergency surgery. Myocardial injury after non-cardiac surgery (MINS) is a frequent but often unrecognized postoperative complication. MINS is associated with an increased risk of other cardiac complications and 30-day mortality. However, the literature on MINS is mainly regarding patients undergoing a wide range of elective or acute surgical procedures, and we do not know if the dynamic TnI-criteria used for acute myocardial injury has any association with mortality in patients with MINS.

This study aims to estimate the incidence of MINS in patients undergoing AHA surgery, and the association between the short-term mortality and MINS defined as a single increased measurement of TnI and as TnI dynamics respectively.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients undergoing acute high-risk abdominal surgery

Exclusion Criteria:

* Patients with microscopic perforations in colonic diverticulitis managed with laparoscopic lavage or drainage
* If further treatment postoperatively was assessed as futile and terminated immediately after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for gastrointestinal perforation, obstruction due to volvulus, tumour, strangulated hernia or adhesions, mesenterial ischemia or necrosis, or anastomotic leakage after gastrointestinal surgery.
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The incidence of MINS within the first four postoperative days | The first four postoperative days
  Postoperative troponin I level equal to or above 59 ng/L

SECONDARY OUTCOMES:
The incidence of dynamic plasma Troponin I changes | The first four postoperative days
  Patients with postoperative troponin I level equal to or above 59 ng/L and a change of +20%

OTHER OUTCOMES:
The association between MINS and all-course mortality within 30 days, 90 days, and 1 year | 30-day, 90-day and 1-year
  MINS defined as troponin I equal to or above 59 ng/L and mortality as yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Bertelsen, Study Chair — Nordsjaellands Hospital
Locations (1):
- Copenhagen University Hospital - North Zealand, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kanstrup CTB, Serup CM, Svarre KJ, Rasmussen MC, Lundstrom LH, Kleif J, Bertelsen CA. Association between troponin I levels and mortality among patients undergoing acute high-risk abdominal surgery-A cohort study. World J Surg. 2024 Feb;48(2):361-370. doi: 10.1002/wjs.12035. Epub 2024 Jan 12. PMID 38284768